CLINICAL TRIAL: NCT04931264
Title: Validation of the YuWell YE660D Oscillometric Upper-arm Blood Pressure Monitor for Clinic and Home in General Population According to the AAMI/ESH/ISO Universal Standard (ISO 81060-2:2018)
Brief Title: Clinical Trial of YuWell YE660D Blood Pressure Monitor in General Population According to the ISO 81060-2:2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Jiangsu Yuyue medical equipment & supply Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, zhang Hui Jie, Director of Clinical Trial Center, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: YUWELL-YLQX202101
Record Dates: First submitted 2021-06-12; First posted 2021-06-18 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Blood Pressure
Keywords: blood pressure monitor; blood pressure measurement; validation study; AAMI/ESH/ISO Universal Standard; ISO 81060-2:2018; YuWell YE660D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YuWell YE660D and mercury sphygmomanometer (Experimental): Blood Pressure Measurement with the YuWell YE660D Electronic Sphygmomanometer (YuWell YE660D) and with Desk Mercury Sphygmomanometer.
  Interventions: Diagnostic Test: YuWell YE660D Electronic Sphygmomanometer

INTERVENTIONS:
Diagnostic Test: YuWell YE660D Electronic Sphygmomanometer — Measurement blood pressure by YuWell YE660D Electronic Sphygmomanometer and Desk Mercury Sphygmomanometer

SUMMARY:
The purpose of this study is to evaluate the accuracy of the YuWell YE660D oscillometric upper-arm blood pressure monitor for clinic and home in general population according to the Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO) Universal Standard (ISO 81060-2:2018).

ELIGIBILITY:
Inclusion Criteria:

* 12 Years and older;
* Subjects voluntarily participate in the clinical trial and sign the informed consent.

Exclusion Criteria:

* Disturbance of consciousness;
* Patients requiring hemodialysis;
* Taking anticoagulant drugs due to cardiovascular and cerebrovascular diseases;
* Pregnant and lactating women;
* Patients with cardiac arrhythmias;
* Other conditions that the investigator considers ineligible for clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurement data | 30 minutes
  Systolic Pressure and Diastolic Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Long, MD，PHD, Study Director — The Second Hospital of Nanjing Medical University
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No